CLINICAL TRIAL: NCT04523974
Title: Preemptive Surgical Intervention and Precise Efficacy Evaluation for Hyperparathyroidism Secondary to Chronic Kidney Disease
Brief Title: Preemptive and Precise Intervention for CKD-SHPT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Bo Shen, Attending Physician, Shanghai Zhongshan Hospital
Other Study IDs: PP-CKD-SHPT
Record Dates: First submitted 2020-08-17; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Hyperparathyroidism; Secondary, Renal
MeSH Terms: conditions — Hyperparathyroidism; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples will be collected to evaluate the level of immunoreactive parathyroid hormone, 25(OH)Vitamin D, calcium, phosphate, alkaline phosphatase and biomarker series of osteogenic collagen metabolism and transformation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preemptive and Precise Intervention: Preemptive surgical intervention will be performed on enrolled CKD-SHPT patients. Safety and efficacy of this intervention will be evaluated during peri-operative period, and long-term outcomes will be analyzed during 1-year follow-up.
  Interventions: Procedure: Preemptive Surgical Intervention and Precise Efficacy Evaluation of CKD-SHPT

INTERVENTIONS:
Procedure: Preemptive Surgical Intervention and Precise Efficacy Evaluation of CKD-SHPT — 1. Preemptive surgical intervention for CKD-SHPT patients with poor calcium and phosphorus metabolism controlled by drugs;
  2. Rapid immunoreactive parathyroid hormone detection technology during peri-operative period.

SUMMARY:
Through multi-center randomized controlled trial studies on preemptive surgical intervention in patients with chronic kidney disease (CKD) - secondary hyperparathyroidism (SHPT), to precisely evaluate the safety and effectiveness during perioperative period, and the long-term outcomes by 1-year follow-up. The follow-ups include the evaluation of the overall quality of life, calcium and phosphorus metabolism, hyperparathyroidism level, vitamin D metabolism, bone mineral density, soft tissue and vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* 1) Chronic Kidney Disease Stage 3-5d patients aged ≥18 years;
* 2) The diagnosis is consistent with CKD-metabolic bone disease and SHPT after evaluation by a kidney specialist;
* 3) Sustained blood immunoreactive parathyroid hormone level of > 300ng/ml, and had received drug treatment;
* 4) Persistent hypercalcemia and/or hyperphosphatemia that is not responding to medication;
* 5) Imaging suggested evidence of at least one parathyroid nodular hyperplasia;
* 6) Signed the informed consent.

Exclusion Criteria:

* 1) Age <18 years old;
* 2) Patients with dialysis duration < 3 months, or with other unstable dialysis state;
* 3) Kidney transplant patients;
* 4) Who is considered inappropriate to participate in this study after evaluation by the supervising physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD 3-5d patients with the diagnosis of CKD-metabolic bone disease and SHPT, with sustained blood immunoreactive parathyroid hormone level of > 300ng/ml, and persistent hypercalcemia and/or hyperphosphatemia, which are not responding to medication.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of preemptive surgical intervention | October 2020 to September 2022
  The rate of post operative complications(including bleeding, infection, adjacent tissue injury) of early precise parathyroidectomy surgery in patients with CKD-SHPT, according to the electronic medical records of the hospital.
Efficacy of preemptive surgical intervention | October 2020 to September 2022
  The rate of relapse of hyperparathyroidism after parathyroidectomy, according to the immunoreactive parathyroid hormone concentration.

SECONDARY OUTCOMES:
short-term and long-term mortality | October 2020 to September 2022
  The all-cause mortality rate and cardiovascular and cerebrovascular mortality rate during hospitalization, by Day 60, Day 180 and 1 year during follow-up.
short-term and long-term bone metabolism | October 2020 to September 2022
  The level of immunoreactive parathyroid hormone, 25(OH)-vitamin D, calcium, phosphate, alkaline phosphatase and biomarker series of bone metabolism during hospitalization, by Day 60, Day 180 and 1 year.
Medical Outcomes Short-Form Health Survey (SF36) Scale | October 2020 to September 2022
  Medical Outcomes Short-Form Health Survey (SF36) scale on quality of life during hospitalization, by Day 60, Day 180 and 1 year during follow-ups. The minimum value is 0, and the maximum value is 100, and higher scores mean a better outcome.
cardiovascular function | October 2020 to September 2022
  The left ventricular ejection fraction (%, obtained by echocardiography) during hospitalization, by Day 180 and 1 year during medical visits.
inpatient days | October 2020 to September 2022
  Length of hospitalization, according the electronic medical records.
hospitalization costs | October 2020 to September 2022
  Cost of hospitalization, according the electronic medical records.
adverse events associated with metabolic bone disease | October 2020 to September 2022
  e.g. fall down, bone fracture during follow-ups, through medical visits and telephone follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Shen, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No